CLINICAL TRIAL: NCT00216827
Title: Calcipotriol Plus Betamethasone Dipropionate Gel Compared to Betamethasone Dipropionate in the Gel Vehicle, Calcipotriol in the Gel Vehicle, and the Gel Vehicle Alone in Scalp Psoriasis
Brief Title: Efficacy and Safety of Calcipotriol Plus Betamethasone Gel in the Treatment of Scalp Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBL 0405 INT
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis of Scalp
MeSH Terms: interventions — calcipotriene; betamethasone-17,21-dipropionate

INTERVENTIONS:
Drug: Calcipotriol plus betamethasone dipropionate (LEO80185 gel)

SUMMARY:
The purpose of this study is to evaluate whether once daily treatment for up to 8 weeks of calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate) gel is safe and more effective than betamethasone 0.5 mg/g (as dipropionate) in the gel vehicle, calcipotriol 50 mcg/g in the gel vehicle or the gel vehicle used alone in patients with scalp psoriasis.

The primary outcome is the proportion of patients with absence of disease or very mild disease after 8 weeks of treatment.

ELIGIBILITY:
Main Inclusion Criteria:

* Scalp psoriasis amenable to topical treatment
* Psoriasis vulgaris on trunk and/or limbs
* Extent of scalp psoriasis involving more than 10% of the total scalp area
* Disease severity on the scalp graded as mild or worse by the investigator
* Consenting out-patients of 18 years or above

Main Exclusion Criteria:

* PUVA or Grenz ray therapy within 4 weeks prior to randomisation
* UVB therapy within 2 weeks prior to randomisation
* Systematic treatment with biological therapies, with a possible effect on scalp psoriasis within 6 months prior to randomisation
* Systemic treatment with all other therapies than biologicals, with a possible effect on scalp psoriasis (e.g., corticosteroids, vitamin D analogues, retinoids, immunosuppressants) within 4 weeks prior to randomisation
* Any topical treatment of the scalp (except for medicated shampoos and emollients) within 2 weeks prior to randomisation
* Topical treatment of the face, trunk and/or limbs with very potent WHO group IV corticosteroids within 2 weeks prior to randomisation
* Current diagnosis of erythrodermic, exfoliative or pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1485
Dates: Start 2004-11; Study Completion 2005-09

PRIMARY OUTCOMES:
Overall disease severity according to investigator's assessment at week 8

SECONDARY OUTCOMES:
Total sign score at week 8
Score for scaliness, redness and thickness at week 8
Extent of scalp psoriasis at week 8
Overall disease severity according to investigator's assessment at week 2 and 4
Overall disease severity according to patients at week 8
Adverse events
Laboratory data

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Jemec, MD, Principal Investigator — Roskilde Hospital, Division of Dermatology
Locations (8):
- FRCPC, Centre de Recherche Dermatologique du Quebec Metropolitain, Québec, Canada
- Roskilde Hospital, Division of Dermatology, Roskilde, Denmark
- Hôpital de l'Archet, Service de Dermatologie, Nice, France
- Hudlegekontoret, Sandvika, Norway
- Hospitais da Universidade de Coimbra, Servico de dermatologia, Coimbra, Portugal
- Hospital Virgen de la Macarena, Servicio de Dermatología, Seville, Spain
- Akademiska Sjukhuset, Hudkliniken, Uppsala, Sweden
- Western Infirmary, Dermatology Department, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en